CLINICAL TRIAL: NCT04404543
Title: A Phase I, Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics and Clinical Activity of SYHA1807 Given Orally in Subjects With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of SYHA1807 in Subjects With Extensive-Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1807-CSP-001
Record Dates: First submitted 2020-05-14; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escalation Cohort (Experimental): Five dose levels will be tested according to the "3 + 3" dose-escalation design.
  The dose-limiting toxicity (DLT) will be assessed from the first administration of SYHA1807 to the end of the first cycle (28 days).
  Interventions: Drug: SYHA1807
- Dose Expansion Cohort (Experimental): Once the RP2D has been determined, an expansion cohort of up to 12~40 subjects will be enrolled in order to better characterize the clinical activity and safety profile of the RP2D.
  Interventions: Drug: SYHA1807

INTERVENTIONS:
Drug: SYHA1807 — Escalation Cohort Administration: Orally
  Arms: Escalation Cohort
Drug: SYHA1807 — Dose Expansion Cohort Administration: Orally
  Arms: Dose Expansion Cohort

SUMMARY:
This is a phase I, open-label, multi-center, non-randomized, 2-part first time inhuman (FTIH) study for SYHA1807. Part 1 is a dose escalation phase to determine the recommended phase 2 dose (RP2D) for SYHA1807 based on the safety, tolerability and pharmacokinetics (PK) profiles observed after oral administration of SYHA1807. The dose escalation study will be performed according to the 3+3 design. Once RP2D is identified, an expansion cohort (Part 2) of up to 12~40 subjects will be enrolled to further evaluate the clinical activity and tolerability of SYHA1807 in subjects with extensive-stage Small Cell Lung Cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced SCLC;
* ECOG(Eastern Cooperative Oncology Group) performance status of 0 or 1;
* Measurable disease according to RECIST v1.1;
* Recovered from all toxicities associated with previous treatments;
* Life expectancy ≥ 3 months;
* Adequate organ function;
* Use of reliable contraceptive methods;
* Signed informed consent from the patient;

Exclusion Criteria:

* Patients with primary malignant tumor other than small cell lung cancer;
* Identified central nervous system metastasis (such as brain metastasis or meningeal metastasis);
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Inadequate washout period for previous anti-tumor therapy;
* Previous treatment with any LSD1(lysine specific demethylase 1) inhibitor;
* Unable to swallow oral medications;
* History of serious systemic diseases;
* History of serious autoimmune diseases；
* HIV positive;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1:Number of Participants With Adverse Events | Through study completion, an average of 2 year
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Part 1:Number of Participants With Serious Adverse Events (SAEs) | Through study completion, an average of 2 year
  SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/birth defect, other situations and is associated with liver injury or impaired liver function.
Part 1:Number of Participants With Dose Limiting Toxicities (DLT) | Through study completion, an average of 2 year
  An event was considered a DLT if it occurs within the first 28 days of treatment.
Number of Participants With Dose Reduction or Delays | Through study completion, an average of 2 year
  The number of participants who had any dose reduction or delay have been presented. All dose reductions were due to AEs.
Number of Participants Withdrawn Due to Toxicities | Through study completion, an average of 2 year
  Participants were monitored from start of the study till the development of toxicity. The data for number of participants withdrawn due to toxicities has been presented.
Number of Participants With Change in Clinical Chemistry Toxicity Grade From Baseline | Through study completion, an average of 2 year
  Baseline value was defined as the most recent, non-missing value from a central laboratory prior to or on the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The number of participants with any grade increase in hematology parameters have been presented.
Number of Participants With Critical Changes in Values of Vital Signs in Response to Drug | Through study completion, an average of 2 year
  Vital sign measurements includes systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature, respiration rate and heart rate. The number of participants with critical changes in values of vital signs in response to drug have been presented.

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) Following Single Dose Administration of SYHA1807 | Through study completion, an average of 2 year
  The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed.
Maximum Observed Plasma Concentration (Cmax) Following Single and Repeat Dose Administration of SYHA1807 | Through study completion, an average of 2 year
  The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed.
Time to Reach Cmax (Tmax) Following Single and Repeat Dose Administration of SYHA1807 | Through study completion, an average of 2 year
  The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed. Tmax is the time to reach Cmax, determined directly from the concentration-time data.
Apparent Terminal Phase Elimination Rate Constant (λz) Following Single and Repeat Dose Administration of SYHA1807 | Through study completion, an average of 2 year
  The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed.
Apparent Terminal Phase Half-life (T1/2) Following Single and Repeat Dose Administration of SYH1A1807 | Through study completion, an average of 2 year
  The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed.
Number of Participants Achieving Disease Control Rate at Week 6、12 | Through study completion, an average of 2 year
  Clinical response was assessed by the investigator using computer tomography or magnetic resonance imaging scans. Clinical response was defined as disease control rate ,CR(Complete response)+PR(Partial response)+SD(Stable disease),based on RECIST version 1.1 at Week 6、12.

OTHER OUTCOMES:
Value of NSE(Neurospecific enolase)、Pro-GRP(pro-gastrin releasing peptide)、CT (calcitonin) With Change From Baseline | Through study completion, an average of 2 year
  Analysis of the relationship between NSE(Neurospecific enolase)、Pro-GRP(pro-gastrin releasing peptide)、CT (calcitonin) NSE and anti-tumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Lou, Study Chair — Department of Medicine, CSPC Clinical Development Division